CLINICAL TRIAL: NCT04292964
Title: Prognostic Factors of Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Clinical Professor, Chongqing Medical University
Other Study IDs: 2020-02-2
Record Dates: First submitted 2020-03-01; First posted 2020-03-03 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: SARS-CoV-2; Outcome, Fatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The outbreak of coronavirus disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in China has been declared a public health emergency of international concern. Despite lower mortality rate, SARS-CoV-2 has killed more people than SARS and MERS and the number keeps growing. Epidemic studies have been well described clinical features of patients with COVID-19, with the disease severity being an independent predictor of poor outcome. However, there is still no research investigating the prognostic factors of patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged >=18years old;
* Diagnosed with CONVID19. Diagnostic criteria including: Laboratory (RT-PCR) confirmed SARS-Cov-2 infection; CT of the lung conformed to the manifestation of viral pneumonia.
* Criteria for severe or critical ill conditions: Respiratory rate >=30/min; or Rest SPO2<=93%; or PaO2/FiO2<=300mmHg.

Exclusion Criteria:

* Near-death state (expected survival time less than 24 hours);
* Malignant tumor;
* Pregnancy or puerperium women;
* Patients who refused to participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
all-cause mortality | 30 days

SECONDARY OUTCOMES:
all-cause mortality | 15 days
Severe state | 15 days
  Criteria for severe or critical ill conditions: Respiratory rate >=30/min; or Rest SPO2<=93%; or PaO2/FiO2<=300mmHg.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wen XS, Jiang D, Gao L, Zhou JZ, Xiao J, Cheng XC, He B, Chen Y, Lei P, Tan XW, Qin S, Zhang DY. Clinical characteristics and predictive value of lower CD4+T cell level in patients with moderate and severe COVID-19: a multicenter retrospective study. BMC Infect Dis. 2021 Jan 12;21(1):57. doi: 10.1186/s12879-020-05741-w. PMID 33435865
- [Derived] Gao L, Jiang D, Wen XS, Cheng XC, Sun M, He B, You LN, Lei P, Tan XW, Qin S, Cai GQ, Zhang DY. Prognostic value of NT-proBNP in patients with severe COVID-19. Respir Res. 2020 Apr 15;21(1):83. doi: 10.1186/s12931-020-01352-w. PMID 32293449